CLINICAL TRIAL: NCT05382676
Title: Prospective Clinical Trials to Assess Performance and Safety of EyeSwift Pro for Assessment of Ocular and Visual Functions
Brief Title: Prospective Clinical Trials to Assess Performance and Safety of EyeSwift Pro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NovaSight (Industry)
Responsible Party: Sponsor
Other Study IDs: NS-00921
Record Dates: First submitted 2022-04-25; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Visual Functions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Visual Function: automated vision measured by EyeSwift®Pro-ESP100
  Interventions: Device: Eyeswift Pro

INTERVENTIONS:
Device: Eyeswift Pro — assessment of visual function parameters

SUMMARY:
EyeSwift Pro assessment of visual function parameters as measured by psychophysics

DETAILED DESCRIPTION:
The following assessments and procedures will be carried out in this trial:

* Baseline assessments will include the following: age, gender, ethnicity, race, education, clinical ocular diagnosis, and general health and use of any concomitant medications.
* Visual and ocular assessment will include unitary testing methods, using the EyeSwift Pro system and the reference method (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* ≥4 years
* Have visual acuity better than 6/60
* Diagnosed as having either Orthophoria or/and Heterophoria or/and Orthotropia or/and heterotopia (group A only)
* Normal vision or visual impermeant (group C and E only)
* Normal or deficient vergence (group D only)
* Normal or deficient reading disabilities (group F only)
* 8 years and older or third grade (group F only)
* Subject in general good health and able, as per investigator decision, to comply with study visits and protocol procedures
* Signed and dated informed consent form
* Parent and participant understand and are willing to comply with

Exclusion Criteria:

* Anophthalmic
* Photosensitive epilepsy or susceptible to epileptic seizures
* Pre-existing concomitant pathology such as congenital cataracts or glaucoma (not including group E)
* Severe developmental delay that would interfere with testing (in the opinion of the investigator). Subjects with mild speech delay or reading and/or learning disabilities are not excluded
* Extraocular muscle (EOM) paralysis (groups A and B only)
* Nystagmus
* Any ocular pathology or anomalies which can interfere with eye-tracking
* Any ocular pathology or anomalies (i.e., age-related macular degeneration (AMD), diabetic retinopathy etc.) (relevant for groups A-F, group E can include such anomalies)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The EyeSwift® Pro-ESP100 is indicated for use in patients aged 3 years and above who are responsive to taking direction and who can pay attention for the duration of the required tests/ protocols
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Automated measurement of heterophoria and heterotropia and detection of a deviating eye in the primary eye position

SECONDARY OUTCOMES:
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Automated measurement of dichoptic divergence and convergence
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Automated measurement of dynamic resolution acuity
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Manual measurement of visual acuity
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Automated measurement of contrast sensitivity
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Presentation of a Worth 4-dot test
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Manual testing of color vision impairments
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Manual measurement of stereoacuity
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Automated analysis of reading patterns
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Automated measurement of fixation stability
measurement by the EyeSwift®Pro-ESP100 | 1 day
  Automated measurement of extraocular motility